CLINICAL TRIAL: NCT01476085
Title: An Open-label Study to Evaluate the Utility of the Apoptosis Imaging Biomarker 18F]ML10 to Assess the Response to Chemotherapy in Patients With Non-Hodgkin's Lymphoma(NHL).
Brief Title: Evaluating the Utility of the Apoptosis Imaging Biomarker 18F]ML10 in Patients With Non-Hodgkin's Lymphoma(NHL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated as ongoing analysis suggested objectives not practical to achieve with study as implemented
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 114238
Record Dates: First submitted 2011-09-01; First posted 2011-11-22 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- no treatment (No Intervention): no treatment
  Interventions: Radiation: ML10

INTERVENTIONS:
Radiation: ML10 — [18F]ML10 radioligand apoptosis biomarker

SUMMARY:
This study aims to evaluate the potential of 2-(5- Fluoro pentyl)-2-methyl malonic acid ([18F]ML10), as an apoptosis imaging biomarker and its potential to predict response in patients with Non Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
Apoptosis or programmed cell death mechanisms are disrupted in cancer cells allowing them to live longer and grow faster than normal cells. Apoptosis is a key target for several novel anti-cancer agents. A biomarker that could permit imaging levels of ongoing apoptosis could be a powerful tool in associated drug development programs by providing relevant data to support proof of concept. In addition, use in the clinical setting may permit the tailoring of treatment for individual patients balancing efficacy of treatment with known toxicity levels. This study aims to evaluate the potential of 2-(5- Fluoro pentyl)-2-methyl malonic acid ([18F]ML10), as an apoptosis imaging biomarker and its potential to predict response in patients with Non Hodgkin's Lymphoma. All patients will have a baseline [18F]ML10 PET-CT scan and a post-treatment scan after the initiation of the first course of intravenous chemotherapy. The study aims to enrol unto 16 subjects with Non-Hodgkins Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent, and willing and able to comply with the requirements and restrictions listed in the consent form.
2. Male or female patients >18 years of age at screening with histological or cytological diagnosis of Non-Hodgkin's Lymphoma and due to receive intravenous chemotherapy for the first time
3. A female subject is eligible to participate if she has non-childbearing potential
4. Male subject must agree to use one of the contraception methods listed
5. Able to lie comfortably on back for up to 70 minutes at a time.
6. WHO performance status 0, 1 or 2 -

Exclusion Criteria:

1. Patients with known history of Hepatitis B, C, non-A, non-B and HIV
2. Any clinically significant medical conditions that in the opinion of the investigator would compromise the compliance with study procedures.
3. Pregnant or breast feeding females.
4. Any other prior anticancer therapy
5. Any new investigational agent, including an investigational anti-cancer agent
6. History of sensitivity to heparin or heparin-induced thrombocytopenia.
7. Males and females not able to comply with contraceptive guidelines during the study.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
changes in [18F]ML10 uptake in tumours | between baseline at day 0 and between 14-20 days after
  Extent of changes in [18F]ML10 uptake in tumours following chemotherapy using visual and semi-quantitative parameters.

SECONDARY OUTCOMES:
alterations in [18F]ML10 uptake with tumour volume and tumour metabolic changes | between baseline at day 0 and between 14-20 days after
  Relationship between alterations in [18F]ML10 uptake with tumour volume and tumour metabolic changes in response to chemotherapy as measured by standard of care CT scan and FDG PET scan.
voxel-based uptake map of [18F]ML10 in the target lesion | between baseline at day 0 and between 14-20 days after
  Alterations in the voxel-based uptake map of [18F]ML10 in the target lesion in response to the chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, London, United Kingdom